CLINICAL TRIAL: NCT06068673
Title: The Potential Impact of Clindamycin on Neurosurgery Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Associate Professor, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Clindamycin in neurosurgery
Record Dates: First submitted 2023-09-29; First posted 2023-10-05 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Neurologic Complication; Neurosurgery
MeSH Terms: interventions — Clindamycin

STUDY DESIGN:
Intervention Model Description: All enrolled 44 patients will be divided into two groups; Group I are patients who will receive clindamycin added-on therapy. Group II patients will be managed with the standard regimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group I are patients who will receive clindamycin added-on therapy.
  Interventions: Drug: Clindamycin 600 mg
- Group B (Active Comparator): Group II patients will be managed with the standard regimen.
  Interventions: Drug: standard regimen

INTERVENTIONS:
Drug: Clindamycin 600 mg — Clindamycin 900 - 1200 mg TWICE per day during 2 weeks period.
  Other Names: Dalacin 600 mg
  Arms: Group A
Drug: standard regimen — standard regimen
  Other Names: Placebo
  Arms: Group B

SUMMARY:
A prospective, open-label, single center, controlled trial. 44 patients that underwent neurosurgery or presented meningitis signs, for whom Clindamycin add-on therapy to assess its effect on neurological complication in relation to Neuron-specific enolase (NSE) and Neurotensin biomarkers levels.

DETAILED DESCRIPTION:
1. This is a prospective, open-label, single center, controlled trial. 44 patients that underwent neurosurgery or presented meningitis signs, for whom Clindamycin add-on therapy is prescribed (900 - 1200 mg twice daily) will be recruited from Alexandria University Main Hospital.
2. Whole blood samples will be collected for Analyses of Neuron-specific enolase (NSE) and Neurotensin will be detected by ELISA.
3. All patients will be assessed for complete blood count (CBC), kidney function, liver function, Methodology

   * Patients will be enrolled if they underwent surgery or presented with clinical signs of meningitis.
   * All enrolled 44 patients will be divided into two groups; Group I are patients who will receive clindamycin added-on therapy. Group II patients will be managed with the standard regimen.
   * Complete physical, laboratory, and radiological assessment will be done for all patients
   * All patients will be followed up during 2 weeks period.
   * Serum samples will be collected for measuring the biomarkers.

ELIGIBILITY:
Inclusion criteria

1) Adult patients will be enrolled if they underwent neurosurgery or presented with clinical signs of meningitis.

Exclusion criteria

1. Age lower than 18.
2. Females with a positive pregnancy test.
3. Known congestive heart failure or ischemic heart disease.
4. Any injury that disturbs the examination (high cervical cord injury or locked-in syndrome, could be a source of bias).
5. Severe brain disease (For example CVA history or brain tumor).
6. Renal failure with GFR lower than 60 ml/min.
7. Patients with unknown identity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Neuron-specific enolase (NSE) Blood Concentration | 2 weeks
  Serum Level of NSE pg/ml
Neurotensin Blood Concentration | 2 Weeks
  Serum Level of Neurotensin pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass Prof., Study Chair — Damanhour University
Locations (1):
- Alexandria University Hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No